CLINICAL TRIAL: NCT03187509
Title: Weight-Based Torsemide Dosing vs. Standard Outpatient Management in Subjects With Heart Failure: A Randomized Open-Label Pilot Study
Brief Title: Weight-Based Torsemide Dosing in Subjects With Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, Robert Siegel, Director of CCU, Jacobi Medical Center, Assistant Professor of Medicine, Albert Einstein College of Medicine, New York City Health and Hospitals Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-7615
Record Dates: First submitted 2017-06-09; First posted 2017-06-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure
Keywords: Torsemide, loop diuretics, weight-based
MeSH Terms: conditions — Heart Failure | interventions — Torsemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weight-Based Torsemide Group (Experimental): Subjects will be randomized to complete a weight-based torsemide dosing regimen for their outpatient heart failure management. These subjects will prescribed a specified dose of torsemide on discharge from the hospital and subsequently have a phone encounter with a physician three times a week where their dose of torsemide will be titrated based on an algorithm which factors in current symptoms and weight. Study subjects will have a final follow-up appointment at the completion of the study to evaluate current symptoms, weight and perform blood work to assess kidney function, electrolytes and brain natriuretic peptide levels.
  Interventions: Drug: Torsemide
- Standard Outpatient Management Group (Active Comparator): Subjects will be randomized to standard outpatient heart failure management where they will be prescribed a fixed daily dose of a loop diuretic upon discharge from the hospital and have a follow-up appointment within one week of discharge. All medications including loop diuretic type, dose and frequency will be managed at the discretion of the patient's primary care physician or cardiologist. Study subjects will have a final follow-up appointment at the completion of the study to evaluate current symptoms, weight and perform blood work to assess kidney function, electrolytes and brain natriuretic peptide levels.
  Interventions: Other: Standard Outpatient Heart Failure Management

INTERVENTIONS:
Drug: Torsemide — These subjects who are randomized to a weight-based torsemide regimen will be instructed via phone encounters three times per week to take an individualized dose of torsemide based on their current weight and symptoms. These subjects will have a follow-up study appointment at week 5 for a final weight and blood work to assess kidney function, electrolytes and brain-natriuretic peptide levels.
  Other Names: Demadex
  Arms: Weight-Based Torsemide Group
Other: Standard Outpatient Heart Failure Management — Those subjects randomized to standard outpatient management group will be prescribed a daily fixed dose of a loop diuretic upon discharge from the hospital. These subjects will have a follow-up appointment within one week of discharge where all medications including loop diuretic type, dose and frequency will be managed at the discretion of the subject's physician. These subjects will also have a follow-up study appointment at week 5 for a final weight and blood work to assess kidney function, electrolytes and brain-natriuretic peptide levels.
  Arms: Standard Outpatient Management Group

SUMMARY:
This study will be a randomized open-label pilot study. The purpose of the study is to compare standard of care outpatient heart failure management versus a weight based torsemide regimen. Subjects admitted to the hospital for heart failure exacerbation will be randomized upon discharge to either standard of care outpatient heart failure management or a weight based torsemide regimen. Those subjects randomized to standard of care therapy will be prescribed a daily fixed dose of a loop diuretic at hospital discharge and have a follow-up appointment within one week of discharge. All management decisions including loop diuretic type, dose and frequency will be made at the discretion of the subject's personal physician. Those randomized to an individualized weight based torsemide regimen will be prescribed a dose of torsemide upon hospital discharge based on a prespecified algorithm. These subjects will then undergo physician-subject phone encounters three times a week where the subject's torsemide dose will be modified based on the prespecified algorithm which incorporates current symptoms and weight. Primary end-point will be an unbiased estimate of 30-day all cause readmission rates. Secondary end-points include incidence of acute kidney injury, changes in brain natriuretic peptide levels from baseline and a preliminary estimate of the effect size and feasibility of a weight-based torsemide regimen intervention in order to plan a future larger study.

DETAILED DESCRIPTION:
This study will be an open-label parallel randomized pilot study comparing an individualized weight-based torsemide dosing regimen vs. standard outpatient management in patients with a diagnosis of heart failure.The study will include consenting subjects who are admitted to Jacobi Medical Center with heart failure and were treated with loop diuretic therapy during hospitalization. Prior to discharge, these subjects will be randomized to one of two groups, either an individualized weight-based torsemide regimen group vs. a standard heart failure management group.

After randomization, all subjects will undergo an initial assessment prior to discharge. All subjects will be examined, weighed and assigned a composite congestion score (CCS). CCS is a measurement of current fluid status that has been shown to correlate with clinical outcomes in heart failure patients (19). It assesses a patient's signs and symptoms of congestion, including dyspnea, orthopnea, fatigue, jugular venous distention, rales and peripheral edema. Each category is given a score from 0-3, 0=none, 1=mild,2=moderate and 3=severe. Each subject is given a final composite score for their current volume status.

After discharge, those randomized to standard care will receive standard heart failure care as currently provided in our institution. This routinely includes, but is not limited to, an appointment with their primary care physician within one week of discharge, nutrition consultation, and social work evaluation with support services provided as determined by the social worker. At discharge, all heart failure medication changes including diuretic type, dose and frequency, as well as further management decisions, will be left to the discretion of the subject and the subject's doctors. Those who will be randomized to the individualized weight-based torsemide regimen will be given a standup home scale and torsemide 20mg tabs in a bottle with 100 tablets.

An initial torsemide dose will be assigned based on the patient's GFR and CCS at discharge. These subjects will then have a phone encounter with a physician three times a week where subjects will be instructed to modify the torsemide dose based on their current weight. Patients will be instructed to weigh themselves at the same time of the day, postvoid, prior to eating, prior to the medication dose, and while wearing the same clothing for consistency. The scales should stand on a flat, solid surface rather than carpets unless specifically designed for use in that setting. All phone call encounters and loop diuretic changes will be based on the pre-specified algorithm. These subjects will also receive all the same care and support as a standard subject, including the primary care appointment in one week and other support services, except with instructions to the subject and provider to follow the loop diuretic recommendations from this protocol. Subjects who have been instructed to take more than 80 torsemide 20mg tablets will receive a delivery of 100 additional torsemide 20mg tablets.

All subjects in the study will have follow up visit at week 5 from discharge date. Total diuretic use during the study period will be assessed and current symptoms/quality of life will be evaluated using the Kansas City Cardiomyopathy Questionnaire. The patient will receive a physical examination including a final weight and calculation of composite congestion score. Serum B-type natriuretic peptide (BNP) will be obtained as well as a basic metabolic panel and serum magnesium level to assess for electrolyte disturbances and changes in kidney function. Intervention group subjects will have a count of the remaining number of torsemide tablets in the bottle of torsemide given to them at discharge. Compliance with the algorithm will be assessed by comparing the number of remaining tablets with the number of tablets prescribed during the study. Subjects whose follow-up visit occurs over 45 days after the date of hospital discharge for the enrollment hospitalization shall be deemed to be late for follow-up. Acute kidney injury (AKI) will be defined as an increase in serum creatinine concentration of 0.3 at the five-week follow-up visit compared to the final serum creatinine level measured during hospitalization. Adherence will be measured by comparing the number of tablets in the subject's torsemide supply to the number of expected tablets in the torsemide supply. Adherence will be defined as a tablet count consistent with the subject having taken 88% or more of the expected torsemide tablets

ELIGIBILITY:
Inclusion Criteria:

1. All subjects with admission diagnosis of heart failure, including heart failure with reduced ejection fraction (HFrEF) or preserved ejection fraction (HFpEF) treated with loop diuretics during hospitalization
2. Must be at least 18 years old at time of enrollment
3. Must have reliable access to a telephone, and be able to speak and understand English or Spanish over a telephone connection

Exclusion Criteria:

1. Any subject who is currently pregnant
2. Any subject with end-stage renal disease requiring hemodialysis
3. Any subject with serum potassium concentration < 3.5 mEq/L at discharge
4. Any subject with serum magnesium concentration < 1.4 mg/dL at discharge
5. Any subject with a known history of allergic reaction to loop diuretics
6. Any subject with known severe stenotic valvular heart disease
7. Any subject who requires chronic inotropic pharmacotherapy
8. Any subject undergoing evaluation for cardiac transplantation or left-ventricular assist device
9. Any subject who is not able to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
30-day all-cause readmission rate | 30 days from enrollment
  To gain an unbiased estimate of 30-day all-cause hospital readmission rate with an individualized weight-based torsemide dosing regimen and with standard therapy

SECONDARY OUTCOMES:
Effect size of weight based torsemide regimen compared to standard therapy | 30 days from enrollment
  To obtain a preliminary estimate of the effect size of an individualized weight-based torsemide regimen intervention using contemporaneous controls of standard care for planning a potential, larger future study
Feasibility of a weight based torsemide regimen | 30 days from enrollment
  To assess the feasibility of subjects to follow an individualized weight-based torsemide regimen as assessed by compliance with study medications, adhering to thrice weekly phone encounters and following medication dose modifications based on the study algorithm. Compliance with the study medication and algorithm will be assessed at the final study appointment by comparing the number of remaining torsemide tablets in the subject's pill box which was provided at the beginning of the study with the number of tablets prescribed during the study.
Incidence of acute kidney injury (AKI) | 30 days from enrollment
  To gain an unbiased estimate of AKI incidence, as defined by an increase serum creatinine by ≥0.3 mg/dL from baseline, with an individualized weight-based torsemide dosing regimen and with standard therapy
Comparison of baseline changes of brain natriuretic peptide (BNP) levels | 30 days from enrollment
  To compare changes in BNP(pg/mL) levels from baseline in subjects randomized to a weight-based torsemide regimen and those randomized to standard therapy

CONTACTS AND LOCATIONS:
Overall Officials: Robert Siegel, MD, Principal Investigator — Jacobi Medical Center, Albert Einstein College of Medicine
Locations (1):
- Jacobi Medical Cent, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No